

# **Statistical Analysis Plan (SAP)**

Transition cAre inteRvention tarGeted to high-risk patiEnts To Reduce rEADmission: A randomized controlled trial

**TARGET-READ phase 2** 

# **Administrative Information**

| Project number: | 706 |
|----------------------------|--------------------------------------|
| Trial registration number: | ID 2018-00084 |
| SAP version: | 1.0, 05.03.2019 |
| Protocol version: | Version 1.1, 13.02.2018 <sup>1</sup> |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|------------|-----------------------------|-------------|
| C TO Belli | Version 1.0 | Page 1 I 27 |



# Authored by

| Name | Affiliation | Role in SAP writing |
|---|---|---|
| Lukas Bütikofer | CTU Bern | Author |
| Andreas Limacher | CTU Bern | Reviewer |
| Jacques Donzé | Médecine interne, Hôpital neuchâtelois | Reviewer |

# **Revision history**

| Revision | Justification | Date |
|----------|-----------------|------------|
| 1.0 | Initial version | 05.03.2019 |

# Approved by

| Name | Affiliation | Study Role | Date and Signature (wet ink) |
|---|---|---|---|
| Lukas Bütikofer | CTU Bern | Trial statistician | |
| Andreas Limacher | CTU Bern | Senior statistician | |
| Jacques Donzé | Médecine interne,<br>Hôpital neuchâtelois | Sponsor-<br>Investigator | |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



b UNIVERSITÄT BERN

# **Contents**

| | CIO Bern | Version 1.0 | Page 3 I 27 |
|---|---|---|---|
| | CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
| | 6.1 | Outcome definition | 19 |
| 6 | Anal | ysis | 19 |
| | 5.6 | Procedural characteristics | 16 |
| | 5.5.3 | 3 Index diagnosis | 15 |
| | 5.5.2 | 2 Index admission and HOSPITAL score | 14 |
| | 5.5.1 | Sociodemographics | 13 |
| | 5.5 | Baseline patient characteristics | 13 |
| | 5.4 | Withdrawal/follow-up | 13 |
| | 5.3 | Recruitment | 13 |
| | 5.2 | Eligibility | 13 |
| | 5.1 | Screening data | 13 |
| 5 | Trial | Population | 13 |
| | 4.4.2 | Per-protocol set (PPS) | 12 |
| | 4.4.1 | Full analysis set (FAS) | 12 |
| | 4.4 | Analysis populations | |
| | 4.3 | Adherence and protocol deviations | |
| | 4.2 | Confidence intervals and p-values | |
| | 4.1 | General | |
| 4 | | stical principles | |
| | 3.2 | Data validation | |
| Ü | 3.1 | Data export | |
| 3 | | ı management | |
| | 2.8 | Blinding | |
| | 2.0 | Timing of final analysis Timing of outcome assessments | |
| | 2.5<br>2.6 | Statistical interim analyses and stopping guidance | |
| | 2.4 | Stratification | |
| | 2.3 | Sample size | |
| | 2.2 | Randomization | |
| | 2.1 | Trial design | |
| 2 | | y methods | |
| | 1.2 | Objectives | 5 |
| | 1.1 | Background and rationale | 5 |
| 1 | Intro | duction | 5 |



#### b UNIVERSITÄT BERN

| 6.1. | .1 Primary outcome | 19 |
|-----------|---------------------------------|----|
| 6.1. | .2 Secondary outcomes | 19 |
| 6.2 | Outcome derivation | 19 |
| 6.3 | Analysis methods | 21 |
| 6.3. | .1 Primary analysis | 21 |
| 6.3. | .2 Secondary analyses | 22 |
| 6.3. | .3 Sensitivity analyses | 22 |
| 6.3.4 | .4 Subgroup analyses | 22 |
| 6.4 | Missing data | 24 |
| 6.4. | .1 Multiple imputations | 24 |
| 6.5 | Evaluation of safety parameters | 25 |
| 6.6 | Statistical software | 25 |
| 6.7 | Quality control | 25 |
| 7 Cha | anges from the protocol | 26 |
| Reference | ces | 27 |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 1 Introduction

# 1.1 Background and rationale

This statistical analysis plan (SAP) serves to describe the methods and time points of the statistical analysis performed for the randomized controlled trial TARGET-READ phase 2 (transition care intervention targeted to high-risk patients to reduce readmission).

### 1.2 Objectives

The primary objective is to evaluate the effect of a transitional care intervention ("TARGET" intervention) prioritized to higher-risk medical patients on the composite of 30-day unplanned readmissions and death.

Secondary objectives are to evaluate:

- the effect of a targeted transitional care intervention to higher-risk medical patients on hospital utilization, medication adherence, patient's perspective on quality of transition of care and time to readmission or death (whatever comes first),
- the effect of a targeted transitional care intervention on the primary outcome in subgroup population of patients with intermediate (simplified HOSPITAL score of 4 or 5) compared to high risk of readmission (simplified HOSPITAL score ≥6), who suffer from common chronic diseases (diabetes, chronic heart failure, COPD or cancer), and according to living place, living status and health insurance,
- the cost-effectiveness of the transitional care intervention.

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 2 Study methods

### 2.1 Trial design

The study is a national multicenter single-blinded randomized controlled trial.

#### 2.2 Randomization

Allocation of patients is done when all inclusion and exclusion criteria are satisfied. Patients are randomly assigned in a ratio of 1:1 to one of two treatment arms:

- 1) Transitional care (intervention) or
- 2) Usual care (control).

Allocation of patients is done with the data management system (REDCap<sup>™</sup>) that also hosts the electronic case report forms (eCRFs). Allocation is stratified by:

- Discharge site (Hôpital Fribourgeois, Centre hospitalier Bienne, CHUV Lausanne, Hôpital neuchâtelois)
- Readmission risk category according to the simplified HOSPITAL score (intermediate vs high risk, i.e. a HOSPITAL score of 4 or 5 vs ≥6)

The readmission risk category is documented on eCRF "Eligibility" by variable <code>strat\_1</code>, the discharge site is coded via the patient ID. The random allocation is performed centrally within the data management system using permuted block with random block sizes of 2, 4 and 6. Investigators receive the allocation only after the eCRF "Eligibility" has been completed. The allocation is documented by variable <code>alloca group</code> on eCRF "Eligibility".

#### 2.3 Sample size

Because we will target patients at higher risk of readmission, we hypothesize that the intervention could reduce the relative risk of readmission by 25%, i.e. more than the 18% reduction found in a recent meta-analysis where patients were mostly not at high risk for readmission. Based on previous findings, the expected 30-day readmission and death rate for patients at intermediate or high risk according to the simplified HOSPITAL score is around 27%. Allowing for 10% loss to follow-up, we determine that we will need 1,380 patients for the study to have 80% power, i.e. 690 in each arm.

The intervention phase (randomized controlled trial) will be restricted to the eligible patients who are at intermediate to high risk of 30-day readmission according to the simplified HOSPITAL score, i.e. ≥4/13 points. We estimate to have around 18,000 patients discharged during the 20-month study period, 30% of which (5,400) will be at higher-risk for a 30-day readmission or death. This should be enough to reach the targeted sample size within the study time frame.

#### 2.4 Stratification

Unless explicitly mentioned, all primary analyses will be stratified for the factors used at randomization (section 2.4).

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 2.5 Statistical interim analyses and stopping guidance

There is no interim analysis planned, i.e. there are no stopping rules on the individual or trial level.

# 2.6 Timing of final analysis

All outcomes will be analyzed collectively after study completion. After completion of data entry, data validation and cleaning will be performed. Data analysis will start after database lock.

# 2.7 Timing of outcome assessments

Table 1: Timing of outcome assessments

| | Index hospitalization <sup>1)</sup> | | Follow-up <sup>2)</sup> (post-discharge) | | |
|---|---|---|---|---|---|
| | Screening<br>(before<br>inclusion) | Visit 1<br>(inclusion, day<br>0) | Visit 2<br>(day3 ±1) | Visit 3<br>(day 14 ±1) | Visit 4<br>(day 30<br>±15) |
| Assessment | Pre-study screening | Baseline and<br>pre- discharge<br>intervention | Post-<br>discharge<br>intervention 1 | Post-<br>discharge<br>intervention 2 | Outcome collection |
| Demography | Χ | | | | |
| Eligibility | Х | | | | |
| HOSPITAL score | Х | | | | |
| Informed consent | | Х | | | |
| Randomization | | Х | | | |
| Baseline characteristics | | Х | | | |
| Medical history | | Х | | | |
| Medication | | Х | | | |
| Activity of daily living (ADL Katz score) | | Х | | | |
| Exposition to intervention | | Х | X | X | |
| Medication discrepancy | | | X | X | |
| Adverse drug event | | | Х | Х | |
| Primary outcome: unplanned readmission or death | | | | | Х |
| Secondary outcomes: | | | | | |
| Number of unplanned readmission | | | | | Х |
| Number of days of hospitalization within 30 days | | | | | Х |
| Diagnoses at readmission or cause of death | | | | | Х |
| Number of emergency department visits | | | | | Х |
| Number of PCP visits | | | | | Х |
| Discharge satisfaction (3-CTM) | | | | | Х |
| Costs of readmission | | | | | Х |

<sup>1)</sup> Assessment based on electronic health record and/or in person.

<sup>2)</sup> Assessment by phone call

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 2.8 Blinding

Most of the study personal including PI, study nurses, statistician and data manager will not be blinded. However, the study nurses collecting the outcomes or working on data cleaning will be blinded to the group allocation.

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 3 Data management

The CRFs in this trial are implemented electronically using a dedicated electronic data capturing (EDC) system (REDCap, https://www.project-redcap.org/). The EDC system is activated for the trial only after successfully passing a formal test procedure. All data entered in the CRFs are stored on a Linux server in a dedicated mySQL database. Responsibility for hosting the EDC system and the database lies with CTU Bern.

# 3.1 Data export

At final analyses, data files will be extracted from the database and imported into a statistical software package according to the SOP for data preparation and programming<sup>2</sup>.

#### 3.2 Data validation

First line data validation is performed by the online eCRF system at real-time as defined in the data dictionary. Second line data validation and cleaning will be performed after completion of data entry but before database lock according to the SOP for data validation<sup>3</sup>.

All baseline characteristics (section 5.5), procedural characteristics (section 5.6) and variables used to derive the outcomes (section 6.2) will be checked for completeness and for outliers. Dates will be checked for consistency (e.g. sequence of date of discharge, intervention phone calls and outcome assessment). The time between discharge and intervention phone calls and outcome assessments will be calculated and values outside the visit windows will be checked.

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|-------------|



# 4 Statistical principles

#### 4.1 General

All recorded and derived variables will be presented by treatment group (and visits, if appropriate) using descriptive summary tables. Continuous variables will be summarized by mean and standard deviation, or median and lower and upper quartiles. Categorical variables will be summarized by absolute and relative frequencies.

In all summaries, the treatment groups will be displayed in the following order: transitional care, usual care. For all parameters, baseline is defined as the last available pre-treatment value (i.e. the last non-missing value available before randomization).

The data collected from patients who are not randomized will only be used for the patient's disposition.

# 4.2 Confidence intervals and p-values

A level of statistical significance of 5% will be used. All statistical testing will be two-sided. All tests will be accompanied by an effect measure (transitional care vs usual care) with a 95% confidence interval (95% CI).

### 4.3 Adherence and protocol deviations

Major protocol deviations are

- Violation of inclusion or exclusion criteria
- · No informed consent signed
- Crossing-over to the other treatment arm
- · Patients not discharged home or to nursing home
- Patients not discharged alive
- Change of HOSPITAL score risk group between inclusion and patient discharge
- Not receiving post-discharge component of the intervention and at least one of the follow-up phone calls (unless the patient was readmitted or died before the follow-up phone call).
- · Blindness breach

These protocol deviations will be summarized by treatment group using absolute and relative frequencies.

Table 2: Derivation of protocol deviations.

| Protocol deviation | eCRF sheet | Variable | Variable type | Derivation |
|---|---|---|---|---|
| Violation of inclusion or excl | Violation of inclusion or exclusion criteria | | | |
| Adult patient | Baseline<br>Characteristics | patient_age | Continuous:<br>years | patient_age<18 |
| Planned discharge home or nursing home | Eligibility | discharged_alive_home | Binary: No, Yes | discharged_alive_home==No |
| Patient expected to be discharged alive? | Eligibility | discharged | Binay: No, Yes | discharged==No |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|------------|-----------------------------|--------------|
| O TO Belli | Version 1.0 | Page 10 I 27 |



| Protocol deviation | eCRF sheet | Variable | Variable type | Derivation |
|---|---|---|---|---|
| Hospital stay of at least<br>24 hours | Baseline<br>Characteristics | computed_nbdays | Continuous:<br>days | computed_nbdays>=1 |
| Patient at higher risk of | Eligibility | hosp_score_simple | Integer: 0-12 | hosp_score_simple<4 |
| 30-day readmission<br>(HOSPITAL score ≥ 4) | Baseline<br>Characteristics | hospital_change<br>hosp_score_simple_2 | Binay: No, Yes<br>Integer: 0-12 | or<br>hospital_change==Yes &<br>hosp_score_simple_2<4 |
| Previous enrolment into the current study | Eligibility | already_enrolled | Binay: No, Yes | already_enrolled==Yes |
| Not living in the country in the next 30 days | Eligibility | home_ch | Binay: No, Yes | home_ch== No |
| No phone to be reached at. | Eligibility | phone | Binay: No, Yes | phone== No |
| Not speaking French or<br>German (depending on<br>the site) | Eligibility | lang | Binay: No, Yes | lang== No |
| Informed consent | Eligibility | consent_signed | Binay: No, Yes | consent_signed==no |
| Crossing-over to the other treatment arm | Protocol<br>Violation | category_interv_notdone<br>category_interv_1funotdone<br>category_interv_2funotdone<br>category_interv_crossover | Binay: No, Yes | (category_interv_notdone==Yes & category_interv_1funotdone==Yes & category_interv_2funotdone==Yes) or category_interv_crossover==Yes |
| Not discharged home or nursing home | Baseline<br>Characteristics | discharged_destination | Categorical: Home, Nursing home, Other acute care Hospital, Acute geriatric, Rehab, Palliative care, Other, Unknown | discharged_destination!=Home<br>&<br>discharged_destination!=Nursing<br>home |
| Not discharged alive | Baseline<br>Characteristics | discharged_alive | Binay: No, Yes | discharged_alive==No |
| | Eligibility | hosp_score_simple | Integer: 0-12 | hospital_change==Yes & |
| Change of HOSPITAL score risk group between | | hospital_change | Binay: No, Yes | hosp_score_simple==4 or 5 & hosp_score_simple_2 > 6 |
| inclusion and patient discharge | Baseline<br>Characteristics | hosp_score_simple_2 | Integer: 0-12 | or<br>hospital_change==Yes &<br>hosp_score_simple>6 &<br>hosp_score_simple_2==4 or 5 |
| Not receiving post-<br>discharge component of<br>the intervention and at | Protocol<br>Violation | category_interv_notdone | Binay: No, Yes | category_interv_notdone==Yes or |
| least one of the follow-up<br>phone calls | Follow-up calls | reach_phone_d3,<br>reach_phone_d14 | Binary: No, Yes | (reach_phone_d3==No & reach_phoned_14==No) |
| Blindness breach | Protocol<br>Violation | description | Free text | Includes "blind" |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



# 4.4 Analysis populations

# 4.4.1 Full analysis set (FAS)

The full analysis set (FAS) will include all randomized subjects. Following the intent-to-treat (ITT) principle, subjects will be analyzed according to the treatment they are assigned to at randomization regardless of the treatment actually received.

# 4.4.2 Per-protocol set (PPS)

The PPS consists of all subjects in the FAS who received the allocated treatment and did not have any major protocol deviations (section 4.3).

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



# 5 Trial Population

# 5.1 Screening data

The number of screened, eligible, consenting and randomized patients will be presented.

# 5.2 Eligibility

Inclusion and exclusion criteria are defined in the study protocol<sup>1</sup>. The number and proportion of patients not fulfilling each criteria will be presented. The reasons for not obtaining an informed consent will be shown.

#### 5.3 Recruitment

A CONSORT patient flow diagram will be drawn following the CONSORT 2010 standards (http://www.consort-statement.org/consort-2010).

### 5.4 Withdrawal/follow-up

All withdrawals and losses to follow-up will be listed with the time points and reasons (if available).

# 5.5 Baseline patient characteristics

Evaluations of the baseline characteristics will be based on the FAS. They will be presented in a descriptive summary table by treatment group—continuous variables as mean and standard deviation or median and quartiles, and categorical variables as absolute and relative frequencies. No statistical comparisons of patient characteristics at baseline will be performed.

#### 5.5.1 Sociodemographics

Sociodemographics are collected on eCRFs "Baseline Characteristics".

Table 3: Sociodemographics.

| Description | Variable | Туре |
|---|---|---|
| Age | patient_age | Continuous: years |
| Gender | gender | Binary: Male, Female |
| Nationality* | nationality | Categorical: Switzerland, Germany,<br>France, Italy, Spain/Portugal, East<br>Europe, Africa, Other, Unknown |
| Living status | living_st | Categorical: With spouse/partner, With another person, Alone, Unknown |
| Living place type* | living_type | Categorical: Home, Protected apartment, Nursing home, Other, Unknown |
| Nurse visits at home† | nurse_home | Categorical: No, Yes, Unknown |
| Support at home for cleaning† | support_home_cleaning | Binary: No, Yes |
| Support at home to buy grocery† | support_home_housing | Binary: No, Yes |
| Support at home for eating† | support_home_eating | Binary: No, Yes |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



| Description | Variable | Туре |
|---|---|---|
| Source of revenue | work | Categorical: Employed, Self-employed,<br>Unemployed, Retired, Invalidity<br>insurance, Social, Other, Unknown |
| Health insurance* | insur | Categorical: Base, Base+compl, Semi-<br>private, Private, Other, No insurance |
| Patient left against medical advice | patient_left | Binary: No, Yes |

<sup>\*</sup>Further specifications are given as free text and will be listed only

# 5.5.2 Index admission and HOSPITAL score

Characteristics of index admission are collected on eCRFs "Baseline Characteristics" and "Costs at Index Diagnoses". Components of the HOSPITAL score are collected on eCRF "Eligibility" and—in case of changes form screening to baseline—on eCRF "Baseline Characteristics".

Table 4: Index admission and HOSPITAL score

| Description | Variable | Туре |
|---|---|---|
| Patient discharged alive | discharged_alive | Binay: No, Yes |
| Destination after discharge* | discharged_destinationr | Categorical: Home, Nursing home, Other acute care Hospital, Acute geriatric, Rehab, Palliative care, Other, Unknown |
| Length of stay | computed_nbdays | Continuous: days |
| Costs (in CHF) of the index hospitalisation | costs_indexhosp | Continuous: CHF |
| HOSPITAL score | | |
| Last hemoglobin level available before discharge | hb_last or hb_last_2† | Continuous: g/l |
| Last sodium level available before discharge | na_last or na_last_2† | Continuous: mmol/l |
| Type of admission | adm_elect or adm_elect_2† | Binary: Elective, Non elective |
| Number of hospitalization at the same hospital in the last 12 months | prevhosp or prevhosp_2† | Integer |
| Length of stay of current hospitalization (in days). | los_index or los_index_2† | Continuous: days |
| Active cancer defined as under treatment, or if remission < 5 years | cancer or cancer_2† | Binay: No, Yes |
| Hospital score (simplified) | hosp_score_simple or<br>hosp_score_simple_2† | Integer 0-12 |

<sup>\*</sup>Further specifications are given as free text and will be listed only

†The former is used if the HOSPITAL score did not change from screening to baseline, the latter if it did change. A change is documented by variable hospital\_change on eCRF "Baseline Characteristics"

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|------------|-----------------------------|--------------|
| C TO Belli | Version 1.0 | Page 14 I 27 |

<sup>†</sup>Not applicable if living type is nursing home



# 5.5.3 Index diagnosis

Information about the index diagnosis is collected on eCRF "Index Diagnosis".

Table 5: Index diagnosis and comorbidities.

| Description | Variable | Туре |
|---|---|---|
| Main diagnosis category* | main_dx_at | Categorical: Heart failure, Acute ischemic heart disease, Arrhythmia, Venous thromboembolism, Stroke/TIA, COPD exacerbation, Pneumonia, Other infection, sepsis, Gastro-intestinal disorder, Liver disorder, Renal disorder, Nutritional or metabolic disorder, Adverse drug event, Neoplasm, Epilepsy, Other |
| Secondary diagnoses and comorbidities* | | |
| Chronic heart failure | comorbidities1 | Binary: Unchecked, Checked |
| Coronary disease | comorbidities2 | Binary: Unchecked, Checked |
| Atrial fibrillation | comorbidities3 | Binary: Unchecked, Checked |
| Peripheral artery disease | comorbidities4 | Binary: Unchecked, Checked |
| Diabetes | comorbidities5 | Binary: Unchecked, Checked |
| Dementia | comorbidities6 | Binary: Unchecked, Checked |
| COPD | comorbidities7 | Binary: Unchecked, Checked |
| Active cancer | comorbidities8 | Binary: Unchecked, Checked |
| Chronic renal failure | comorbidities9 | Binary: Unchecked, Checked |
| Liver cirrhosis | comorbidities10 | Binary: Unchecked, Checked |
| Drug or Alcohol Abuse | comorbidities11 | Binary: Unchecked, Checked |
| Epilepsy | comorbidities12 | Binary: Unchecked, Checked |
| Any treated psychiatric disease | comorbidities13 | Binary: Unchecked, Checked |
| Letter of discharge has been collected | letter_disch_late | Binary: No, Yes |

<sup>\*</sup>Main and secondary diagnoses are also documented as free text (variables main\_dx and dx\_1\_dx20), which will be listed only.

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



#### 5.6 Procedural characteristics

Procedural characteristic include the components of the transitional care intervention and are collected for the transition care group only. The pre-discharge component of the intervention is documented at baseline (visit 1) on eCRF "Pre-discharge component", the follow-up phone calls (visit 2 and visit 3) on eCRFs "Follow-up call 1 (Day 3)" and "Follow-up call 2 (Day 14)". Evaluations of the procedural characteristics will be based on the FAS. They will be presented in a descriptive summary table—continuous variables as mean and standard deviation or median and quartiles and categorical variables as absolute and relative frequencies.

Table 6: Procedural characteristics: pre-discharge components.

| Description | Variable | Type |
|---|---|---|
| <u> </u> | | |
| Basic information about her/his main diseases has been performed? | pat_info | Binary: No, Yes |
| Which information about those comorbidities have been given to the patient? | | |
| Heart failure | inf_shee_giv1 | Binary: Unchecked, Checked |
| Coronary disease | inf_shee_giv2 | Binary: Unchecked, Checked |
| Peripheral artery disease | inf_shee_giv3 | Binary: Unchecked, Checked |
| Atrial fibrillation | inf_shee_giv4 | Binary: Unchecked, Checked |
| Chronic obstructive lung disease | inf_shee_giv5 | Binary: Unchecked, Checked |
| Stroke | inf_shee_giv6 | Binary: Unchecked, Checked |
| Gastrointestinal bleeding | inf_shee_giv7 | Binary: Unchecked, Checked |
| Chronic renal failure | inf_shee_giv8 | Binary: Unchecked, Checked |
| Liver cirrhosis | inf_shee_giv9 | Binary: Unchecked, Checked |
| Thromboembolism | inf_shee_giv12 | Binary: Unchecked, Checked |
| Diabetes | inf_shee_giv13 | Binary: Unchecked, Checked |
| Other* | inf_shee_giv88 | Binary: Unchecked, Checked |
| No listed comorbidity | inf_shee_giv0 | Binary: Unchecked, Checked |
| Medication reconciliation has been performed and explanation about medication list? | med_reco | Binary: No, Yes |
| Have you noticed any medication discrepency that needed to be transmitted to the medical team? | med_reco_disc | Binary: No, Yes |
| Patient education about general health recommendation has been performed? | pat_educ | Binary: No, Yes |
| Dependence Level: score of the Katz Index | katz_ind | Integer: 0-6 |
| Post discharge follow-up visit to the treating physician has been planned?* | folup_plan | Binary: No, Yes |
| Discharge summary sent to the treating physician | dis_sumpcp | Binary: No, Yes |
| Barriers to a safe discharge, including patient's ability to carry out the discharge plan has been assessed | finalcheck | Binary: No, Yes |

<sup>\*</sup>Further specifications are given as free text and will be listed only.

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|----------|-----------------------------|--------------|
| CIOBelli | Version 1.0 | Page 16 I 27 |



Table 7: Procedural characteristics: follow-up call 1 (Day 3) and follow-up call 2 (Day 14).

| Description | Variable | Туре |
|---|---|---|
| Patient reached by phone | reach_phone_d3 or reach_phone_d14† | Binary: No, Yes |
| Reason why the patient wasn't reached* | reas_pat_notre_d3 or<br>reas_pat_notre_d14† | Categorical: Death, No answer,<br>Other |
| Death source of information* | death_sourceinfo_d3 or death_sourceinfo_d14† | Categorical: Next of kin, Treating physician, Hospital, Death certificate, Other |
| Death was due to an accident/trauma? | trauma_death_d3 or<br>trauma_death_d14† | Categorical: No, Yes, Unknown |
| Cause of death (according to certificate of death if possible) | cause_death_d3 or<br>cause_death_d14† | Free text |
| Condition improved since discharge | cond_impr_d3 or<br>cond_impr_d14† | Categorical: No, or rather no, Yes or rather yes, Stable, New symptom |
| Since your discharge of the hospital, do you have more pain? | morepain_d3 or<br>morepain_d14† | Binary: No, Yes |
| How does the mobility/walking distance change since discharge? | red_wal_dis_d3 or<br>red_wal_dis_d14† | Categorical: Mobility/walking distance improved, Mobility/walking remained about the same, Mobility/walking decreased, Not able to evaluate |
| Capacity to prepare meals alone? | cap_meal_d3 or<br>cap_meal_d14† | Binary: No, Yes |
| Weight trend over the last days/weeks | wei_tren_d3 or<br>wei_tren_d14† | Categorical: Increased, Reduced,<br>Stable, Unknown |
| Glucose values most often‡ | glu_val_tre_d3 or<br>glu_val_tre_d14† | Categorical: Between 4-10, >10,<br>Between 10-15, >15, Unkown |
| Do you take your medication as prescribed? | medicasprescribed_d3 or medicasprescribed_d14† | Binary: No, Yes |
| Is there any medication discrepancy between current list and list of discharge? | med_discr_d3 or<br>med_discr_d14† | Binary: No, Yes |
| Presence of any of those medications? | pre_med_d3<br>orpre_med_d14† | Categorical: Anticoagulants,<br>Narcotics and opiates, Sedatives,<br>Insulin |
| Did any of these Adverse Event occur since discharge? | | |
| Dizziness | adv_dru_ev_d31 or<br>adv_dru_ev_d141† | Binary: Unchecked, Checked |
| Bleeding | adv_dru_ev_d32 or<br>adv_dru_ev_d142† | Binary: Unchecked, Checked |
| Hypoglycemia | adv_dru_ev_d33 or<br>adv_dru_ev_d143† | Binary: Unchecked, Checked |
| Delirium | adv_dru_ev_d34 or<br>adv_dru_ev_d144† | Binary: Unchecked, Checked |
| Lethargy / Oversedation | adv_dru_ev_d35 or<br>adv_dru_ev_d145† | Binary: Unchecked, Checked |
| Nausea / vomiting | adv_dru_ev_d36 or<br>adv_dru_ev_d146† | Binary: Unchecked, Checked |
| Fall | adv_dru_ev_d37 or<br>adv_dru_ev_d147† | Binary: Unchecked, Checked |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



| Description | Variable | Туре |
|---|---|---|
| None | adv_dru_ev_d30 or<br>adv_dru_ev_d140† | Binary: Unchecked, Checked |
| Patient had doctor's office visit since discharge | pcp_visit_d3 or<br>pcp_visit_d14† | Categorical: No, Yes as planned,<br>Yes as new appointment |
| Reason why the patient didn't have any treating physician visit since discharge* | reas_no_pcp_d3 or<br>reas_no_pcp_d14† | Categorical: Visit is planned,<br>Patient didn't want/ couldn't,<br>Treating physician couldn't/not<br>available, Other, Unknown |
| Suggestion to see the treating physician was necessary during this follow-up call | sug_see_pcp_d3 or<br>sug_see_pcp_d14† | Binary: No, Yes |
| Patient education about her/his diseases has been refreshed | patient_education_d3 or patient_education_d14† | Binary: No, Yes |

<sup>\*</sup>Further specifications are given as free text and will be listed only

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|

<sup>†</sup>For follow up call 1 and 2, respectively.

<sup>‡</sup>Only for patients with diabetes



# 6 Analysis

#### 6.1 Outcome definition

#### 6.1.1 Primary outcome

The primary outcome is the number of patients who have an unplanned readmission or die within 30 days after discharge.

#### 6.1.2 Secondary outcomes

- Number of deaths within 30 days after discharge
- Number of patients with unplanned readmission within 30 days after discharge
- Time to first unplanned readmission or death within 30 days
- Main cause of readmission or death
- Post-discharge health care utilization within 30 days after discharge from index hospitalization:
  - o number of unplanned hospital readmissions
  - o number of planned hospital readmissions
  - o total number of unplanned days of hospitalizations
  - o total number of planned days of hospitalizations
  - number of emergency room visits
  - o number primary care provider visits
- Patient's perspective (satisfaction) on quality of transition of care between hospital and home assessed by the three-item care transition measure (CTM-3) at 30 days
- Costs of readmission at 30 days

#### 6.2 Outcome derivation

Table 8: Derivation of primary and secondary outcomes.

| Outcome | eCRF sheet | Variable | Variable type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|
| <b>Primary</b> : Unplanned readmission or death within 30 days after discharge | Baseline<br>Characteristics | discharged_alive | Binary: No,<br>Yes | discharged_alive==No<br>or | |
| | Follow-up calls | reas_pat_notre_d3,<br>reas_pat_notre_d14 | Categorical:<br>Death, No<br>answer, Other | reas_pat_notre_d3==Death or reas_pat_notre_d14==Death or death_d30==Yes or unplanned>=1 | Binary |
| | Outcomes 30 | death_d30 | Binary: No,<br>Yes | | |
| | days | unplanned | Integer: 0-6 | | |
| Deaths within 30 days after discharge | Baseline<br>Characteristics | discharged_alive | Binary: No,<br>Yes | discharged_alive==No | |
| | Follow-up calls | reas_pat_notre_d3,<br>reas_pat_notre_d14 | Categorical:<br>Death, No<br>answer, Other | reas_pat_notre_d3==Death<br>or<br>reas_pat_notre_d14==Death | Binary |
| | Outcomes 30<br>days | death_d30 | Binary: No,<br>Yes | or<br>death_d30==Yes | |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



| Outcome | eCRF sheet | Variable | Variable type | Derivation | Outcome<br>type |
|---|---|---|---|---|---|
| Unplanned readmission within 30 days after discharge | Outcomes 30 days | unplanned | Integer: 0-6 | unplanned>=1 | Binary |
| | Baseline<br>Characteristics | disch_date_index,<br>baseline_death | Date: dmy | Time:<br>min(30, min[baseline_death, | |
| Time to first | Follow-up calls | date_death_d3,<br>date_death_d14 | Date: dmy | date_death_d3,<br>date_death_d14,<br>date_death_d30<br>unplanned_in_1,<br>lcontact_date] –<br>disch_date_index) | Time-to-<br>event |
| unplanned<br>readmission or death | Outcomes 30 days | date_death_d30,<br>unplanned_in_1 | Date: dmy | | |
| | End of Study | lcontact_date | Date: dmy | Failure:<br>Primary==Yes | |
| Main cause of | Follow-up calls | cause_death_d3,<br>cause_death_d14 | Free text | Tabulated free text fields will | Categorical |
| readmission or death | Outcomes 30<br>days | dx_read30,<br>cause_death_d30 | Free text | be manually categorized | Categorical |
| Number of unplanned hospital readmissions | Outcomes 30<br>days | unplanned | Integer: 0-6 | - | Count |
| Number of planned hospital readmissions | Outcomes 30 days | planned_readmission | Integer: 0-8 | - | Count |
| Total number of unplanned days of hospitalizations | Outcomes 30 days | unplanned_x_in,<br>unplanned_x_out | Date: dmy | unplanned_x_out –<br>unplanned_x_in | Count |
| Total number of planned days of hospitalizations | Outcomes 30<br>days | tot_rehosp_days_planned | Continuous:<br>days | - | Count |
| Number of emergency room visits | Outcomes 30 days | nb_edvisits | Integer | - | Count |
| Number primary care provider visits | Outcomes 30 days | nb_pcpvisits | Integer | - | Count |
| | Baseline<br>Characteristics | disch_date_index,<br>baseline_death | Date: dmy | min(30, min[baseline death, | |
| Offset for count | Follow-up calls | date_death_d3,<br>date_death_d14 | Date: dmy | date_death_d3,<br>date_death_d14, | Continuous |
| variables | Outcomes 30 days | date_death_d30 | Date: dmy | date_death_d30<br>lcontact_date] –<br>disch_date_index) | |
| | End of Study | lcontact_date | Date: dmy | | |
| Patient's perspective<br>(satisfaction) on<br>quality of transition of<br>care between hospital<br>and home (CTM-3) | Outcomes 30 days | ctm1, ctm2, ctm3 | Binary: No,<br>Yes | ctm1==Yes & ctm2==Yes & ctm3==Yes | Binary |
| Costs of readmission | Costs at<br>Outcomes 30<br>days | costs_30d | Continuous:<br>CHF | - | Continuous |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|-----------|-----------------------------|--------------|



### 6.3 Analysis methods

#### 6.3.1 Primary analysis

The primary analysis will be based on the FAS. Missing data will be handled according to section 6.4.

#### 6.3.1.1 Analysis of the primary outcome

The proportion of patients that have an unplanned readmission or die will be calculated in both groups with a 95% Wilson score confidence interval. For the comparison between the two groups, a Mantel-Haenszel risk difference stratified for the stratification factors used in randomization (section 2.4) will be shown (transitional care – usual care). A two-sided 95% CI will be calculated according to the procedure described by Klingenberg<sup>4</sup>. A stratified Cochran-Mantel-Haenszel test will be used to test for differences (e.g. using emh in Stata).

#### 6.3.1.2 Analysis of secondary outcomes

The number of patients that die will be compared between treatment groups using a Mantel-Haenszel risk difference with a two-sided 95% Cl<sup>4</sup> and a Cochran-Mantel-Haenszel test, both stratified for the stratification factors used in randomization.

The risk of 30 day unplanned readmissions in each group will be estimated using the cumulative incidence function with death as competing event calculated from flexible parametric survival models (e.g. using stpm2 followed by stpm2\_standsurv in Stata)<sup>5,6</sup>. Groups will be compared using the cumulative incidence difference with 95% CI and a z-test, based on delta method standard errors and a normal approximation. We will also report the cumulative incidence of the competing event (death without readmission) for each group and the risk difference between groups.

Time to unplanned readmission or death will be graphically depicted by Kaplan-Meier curves for each treatment group. Groups will be compared using a log-rank test stratified for the stratification factors used in randomization. As an effect measure, we will use the restricted mean survival time truncated at 30 days calculated using flexible parametric survival models with the group and factors used at randomization as covariates<sup>7</sup>. The restricted mean survival time for each group and the difference between groups will be reported with 95% CI and a p-value.

The main cause of readmission or death will mainly be analyzed with descriptive statistics. The number and proportion of patients in each category will be shown for both groups.

Count outcomes (number of hospital readmissions, number of days of hospitalization, number of emergency room visits, number of primary care provider visits) will be presented with number of patients, person-time and incidence rate with 95% CI. Groups will be compared using a negative binomial regression with the group and the stratification factors as covariates and the observation time as offset. An incidence rate ratio with 95% CI and p-value will be reported. In case of an excess of zeros and overdispersion that cannot be modeled by the negative binomial distribution we will consider zero-inflated negative binomial regression (e.g. using function <code>zeroinfl</code> from R package pscl).

Each item of the CTM-3 score will be summarized by treatment group using relative and absolute frequencies. The number of patients with a yes on all items will be compared between treatment groups using a Mantel-Haenszel risk difference with a two-sided 95% Cl<sup>4</sup> and a Cochran-Mantel-Haenszel test, both stratified for the stratification factors used in randomization.

The costs of readmission will be analyzed by linear regression with the treatment group and the stratification factors used in randomization as covariates. The treatment effect will be presented as

| CTU Bern SAP | SAP for TARGET-READ phase 2 | 05.03.2019 |
|--------------|-----------------------------|--------------|



mean difference with 95% CI and a p-value. Model assumption will be checked visually using plots of residuals (residuals vs fitted values, QQ-plot). If model assumptions are violated, transformation of the outcome (e.g. log), more robust methods (e.g. robust standard errors or robust regression) or non-parametric methods (e.g. Wilcoxon-Mann-Whitney test or van Elteren's test) will be considered.

#### 6.3.2 Secondary analyses

All outcomes will also be analyzed in the PPS. Only patients without missing value for the respective outcome will be considered (complete cases).

### 6.3.3 Sensitivity analyses

The following sensitivity analysis will be included for all outcomes:

- 1) Without early readmissions. The primary endpoint will be re-analyzed excluding the patients with unplanned readmissions up to the day after index discharge (i.e. unplanned\_1\_in disch\_date\_index <=1)
- 2) No stratification: All outcomes will be analyzed in crude analyses not adjusting for stratification factors. Binary outcomes will be compared by chis-squared test, continuous outcomes by Student's t-test or the Wilcoxon-Mann-Whitney test, count outcomes using an exact Poissontest and time-to-event outcomes by a log-rank test. Effects will be presented as non-stratified risk difference, mean difference or Mann-Whitney statistic (i.e. the probability that a random patient from the intervention group will have a higher value than a random patient from the control group), incidence rate ratio, and restricted mean survival time difference, respectively, with 95% CI.
- 3) Primary endpoint based on survival methods. The risk of readmission or death at 30 days for both groups and the risk difference between groups will be calculated with 95% CI and p-values from a z-test using a) a flexible parametric survival model for time to unplanned readmission or death with the group and stratification factors as covariates and b) from the Kaplan-Meier-estimator for time to unplanned readmission or death not using the stratification. CIs for the risk differences and the z-test will be calculated using delta method standard errors and a normal approximation.
- 4) Non-parametric unplanned readmissions: The risk of unplanned readmission at 30 days in the presence of the competing risk of death will be calculated for each group using the non-parametric cumulative incidence function estimator with 95% CI according to Choudhury et al<sup>8</sup>. Stratification will be ignored.

#### 6.3.4 Subgroup analyses

The primary outcome will be analyzed for subgroups defined by the stratification factors for randomization:

- Risk for readmission (HOSPITAL score of 4 or 5 vs ≥6)
- Clinical site
- Diabetes
- Chronic heart failure
- COPD
- Cancer

| CTU Bern SAP for TARGET-READ phase 2 Version 1.0 | 05.03.2019 |
|----------------------------------------------------|-------------|
| | Version 1.0 |



- Living place (nursing home vs rest)
- Living status (alone vs rest)
- Health insurance (Semi-private and private vs rest)

Table 9: Derivation of subgroups

| Subgroup | eCRF sheet | Variable | Categorization |
|---|---|---|---|
| | Eligibility | hosp_score_simple | if hospital_change==no: |
| HOSPITAL score | Baseline | hosp_change | hosp_score_simple > 5 else: |
| | Characteristics | hosp_score_simple_2 | hosp_score_simple_2 > 5 |
| Clinical site | - | record_id | substr(record_id,1,3) |
| Diabetes | Index<br>Diagnosis | comorbidities5 | comorbidities5==checked |
| Observator by a set failure | Index | main_dx_at | main_dx_at==Heart failure |
| Chronic heart failure | Diagnosis | comorbidities9 | or<br>comorbidities9==checked |
| 0000 | Index<br>Diagnosis | main_dx_at | main_dx_at==COPD exacerbation |
| COPD | | comorbidities7 | or<br>comorbidities7==checked |
| | Index | main_dx_at | main_dx_at==Neoplasm |
| Cancer | Diagnosis | comorbidities8 | or<br>comorbidities8==checked |
| Living place | living_type | Categorical: Home, Protected apartment, Nursing home, Other, Unknown | living_type==Nursing home |
| Living status | living_st | Categorical: With spouse/partner, With another person, Alone, Unknown | living_st==Alone |
| Health insurance | insur | Categorical: Base,<br>Base+compl, Semi-private,<br>Private, Other, No insurance | insur==Semi-private or insur==Private |

Subgroups will be analyzed using regression models with the treatment group, the subgroup and their interaction and the stratification factors used at randomization as covariates. If possible, a binomial model with identity link function will be used and the effects will be reported as risk differences with 95% Cls. Otherwise, a Poisson model with identity link and robust standard errors (leading to risk differences) or a binomial model with logit link (leading to odds ratios) will be considered. Models with and without interaction will be compared using a likelihood ratio test and the p-value will be reported as p-value for interaction. Results will be presented in a forest plot.

As a secondary analysis, subgroups will be categorized (according to Table 9) and analyzed using Mantel-Haenszel methodology. A risk difference will be shown for each subgroup with both a lower one-sided and a two-sided 95% CI. The p-value from a Mantel-Haenszel test of homogeneity will be presented. The Mantel-Haenszel subgroup analyses will not be stratified for the factors used at randomization.

| CTU Bern SAP for TARGET-READ pha | SAP for TARGET-READ phase 2 | 05.03.2019 |
|---|---|---|
| C TO Belli | Version 1.0 | Page 23 I 27 |



### 6.4 Missing data

The number of patients with non-missing observations will be reported for each outcome.

Missing data may occur due to drop-outs or deaths. The former will lead the absence of all outcome information as outcomes are only assessed once. Since the follow-up is very short we do not expect a lot of drop-outs and it is unlikely that these patients did have a readmission or died. Therefore, we will assume that drop-outs did not have a readmission and did not die. For survival analyses they will be censored at one day. For count outcomes they will be assumed to have no observed event and an offset of one day. For patient satisfaction multiple imputations will be used (section 6.4.1). If the amount of drop-outs is larger than 5%, we will do a sensitivity analysis in which the primary outcome (unplanned readmission or death) will be multiply imputed as a binary variable (section 6.4.1).

Death will not lead to missing data for the primary outcome, 30-day deaths and time to primary outcome. For 30-day unplanned readmission, death is a competing event and the cumulative incidence at 30 days will be used (section 6.3.1.2). Count outcomes will be handled by including the observation time as offset in the Poisson regression. For patient satisfaction multiple imputations will be used (section 6.4.1). In a sensitivity analysis, the worst possible outcome will be assigned to deaths (i.e. a negative respond to all question of the CTM-3).

#### 6.4.1 Multiple imputations

Multiple imputations will be based on the treatment group, and selected baseline and outcome variables (see next section). Since missing values in these variables are possible, chained equations will be used (e.g. with command mi impute chained in Stata). This procedure fills in missing values in multiple variables iteratively based on a sequence of univariate imputation methods with fully conditional specification of prediction equations. Predictive mean matching (pmm) will be used for continuous, logistic regression (logit) for binary and multinomial regression (mlogit) for categorical variables. Survival outcomes will be imputed by adding the log time and the censoring indicator to the imputation model.

Based on such chained equations, a total of 50 multiple imputations will be calculated. If it is not possible to impute all outcomes in one model, a stepwise approach will be considered.

The 50 imputed data sets will be analyzed using Rubin's rules<sup>9</sup> (e.g. with prefix mi estimate in Stata).

#### 6.4.1.1 Selection of variables for multiple imputations

Baseline variable (section 5.5) and outcomes (section 6.1) will be considered for multiple imputations.

Variables with more than 50% missing values will not be used for the imputation model. Binary variables with a frequency of less than 5% in one category will also be omitted. If two binary variables have less than 5% or more than 95% discordant pairs only one of the two will be used (the one with less missings). Levels of ordinal variables with a frequency of less than 5% will be collapsed by adding the entries to the neighbouring category (i.e. next higher or lower level) with the higher frequency (if there are more than one). Categorical variables might generally be recoded if it improves the fit of the imputation model and does not lead to substantial loss of information. Continuous variables will be log-transformed if it improves normality (checked by Shapiro-Wilk tests and QQ plots).

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|----------|-----------------------------|--------------|
| | Version 1.0 | Page 24 I 27 |



From the remaining variables an imputation model will be constructed based on combined clinical and statistical reasoning. All variables that may provide information about the imputed variable will be included.

# 6.5 Evaluation of safety parameters

Since the intervention is of very low risk for the patient safety parameters will not be evaluated.

#### 6.6 Statistical software

The statistical analysis will be performed using the statistical software packages Stata<sup>10</sup> and/or R<sup>11</sup>.

# 6.7 Quality control

A second statistician will reproduce the analysis of the primary outcome (for both the FAS and the PPS) based on the exported data. The risk difference and the 95% confidence interval should not differ by more than 0.01, the p-value by 0.001. Otherwise, the reason for the difference will be determined and a consensus must be reached.

| CTU Bern SAP for TARGET-READ phase 2 Version 1.0 | 05.03.2019 |
|----------------------------------------------------|-------------|
| | Version 1.0 |



# 7 Changes from the protocol

The SAP is consistent with principle features of the statistical methods described in the protocol. The following deviations were made:

Table 10: Changes from protocol

| Header | Change | Reason |
|---|---|---|
| Blinded analysis | Blinded analysis not implemented | The allocation can immediately be seen from the eCRFs because only patients in the intervention group have follow up phone calls. It would therefore need an extra statistician that carefully prepares the data so that it is not possible to see the allocation. Given the open-label nature of the study and the straightforward analysis this additional effort seems not to be justified. |
| Secondary outcome "Medication adherence: 4-item Morisky Medication Adherence Scale (MMAS-4)". | Removed | High license fees would incur |
| Secondary endpoint "Number of planned hospital readmissions" and "Total number of planned days of hospitalizations" | Added | Information about the planned readmissions is of interest but was not considered in the protocol. |
| Test for the analysis of primary and binary secondary outcome | Stratified Cochran-Mantel-Haenszel test instead of simple chi-squared test | Stratification factor should be considered in the analysis |
| Subgroup HOSPITAL score | Categories 4 or 5 vs ≥6 instead of 5 or 6 vs ≥7 | Categories correspond to stratification of the randomization |
| Subgroup clinical site | Added | Used as stratification factor in randomization |
| Subgroups cancer, living place, living status and health insurance | Added | Of interest, not mentioned in protocol |

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|----------|-----------------------------|--------------|
| | Version 1.0 | Page 26 I 27 |



### References

- <sup>1</sup> Clinical trial protocol: Transition care intervention targeted to high-risk patients to reduce readmission (TARGET-READ): A randomized controlled trial, Version 1.1, 13.02.2018
- <sup>2</sup> SOP Data preparation and programming, CS\_STA\_SOP\_05, version 02, 15.08.2015
- <sup>3</sup> SOP Statistical data validation, CS\_STA\_SOP\_02, version 02, 15.08.2015
- <sup>4</sup> Klingenberg, B. 2014. A new and improved confidence interval for the Mantel–Haenszel risk difference. *Statistics in medicine*, 33(17): 2968.
- <sup>5</sup> Royston, P. and Lambert, P.C. 2011. Flexible parametric survival analysis in Stata: Beyond the Cox model. College Station, Texas: Stata
- <sup>6</sup> Hinchliffe, Sally R., and Paul C. Lambert. 2013. "Extending the flexible parametric survival model for competing risks." *The Stata Journal*, 13(2): 344
- <sup>7</sup> Royston, P. and Parmar, M. K. 2013. Restricted mean survival time: an alternative to the hazard ratio for the design and analysis of randomised trials with a time-to-event outcome. *BMC Med Res Methodol*, 13: 152
- <sup>8</sup> Choudhury, Jahar B. 2002. Non-parametric confidence interval estimation for competing risks analysis: application to contraceptive data, *Statistics in medicine*, 21(8): 1129
- <sup>9</sup> Rubin, D. B. 2004. Multiple imputation for nonresponse in surveys. John Wiley & Sons, 81
- <sup>10</sup> StataCorp. 2017. Stata Statistical Software: Release 15. College Station, TX: StataCorp LLC
- <sup>11</sup> R Development Core Team. 2008. R: A language and environment for statistical computing. R Foundation for Statistical Computing. Vienna, Austria

| CTU Bern | SAP for TARGET-READ phase 2 | 05.03.2019 |
|----------|-----------------------------|--------------|
| CTO Bern | Version 1.0 | Page 27 I 27 |